CLINICAL TRIAL: NCT00582062
Title: Detection of Peritoneal Micrometastasis in Gastric and Pancreatic Cancer in Peritoneal Wash Samples
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 06-022
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Gastric and Pancreatic Cancer
Keywords: Gastric Cancer; Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Positive controls will include patients who have positive cytology or positive biopsy of peritoneal metastases. Cell lines which over-express these tumor markers will also be used as positive controls. Sensitivity will be defined using serial dilutions of several established gastric and pancreatic tumor cell lines. The mRNA of the tumor markers will be normalized to glyceraldehyde-3-phosphate dehydrogenase mRNA expression.
  Interventions: Other: washings for experimental marker testing
- 2: Patients who are scheduled to undergo laparoscopy for benign disease (e.g., laparoscopic cholecystectomy, hernia repair, or prophylactic BSO) will be recruited as negative controls. A leukemia cell line which does not express epithelial cell markers will also be used as a negative control for the RT-PCR reactions.
  Interventions: Other: washings for experimental marker testing

INTERVENTIONS:
Other: washings for experimental marker testing — During the laparoscopy, a small amount of a mild salt solution will be introduced to gently wash the inside of the abdomen. The fluid will be removed and sent to the laboratory for two analyses: 1) washings for cytology (routine), and 2) washings for experimental marker testing (experimental).

SUMMARY:
We are undertaking a study of patients with gastric or pancreatic cancer. A common place for cancer to return after surgery for gastric or pancreatic cancer is the inside lining of the abdomen, called "peritoneal metastasis". At the time of surgery, washing the abdomen with a mild salt solution may reveal free cancer cells in the abdomen which could develop into peritoneal metastasis. Recently, surgeons here at Memorial Sloan-Kettering have found that patients who have these cells develop peritoneal metastases and are better treated with chemotherapy rather than surgery. Sometimes, though, these cells might be present but cannot be found by using current techniques. We are trying to figure out a better way to find these free cancer cells. This could improve our treatment of patients with gastric and pancreatic cancer. We need "negative control" population to which we can compare the peritoneal washings of these cancer patients.

DETAILED DESCRIPTION:
Positive peritoneal cytology is a predictor of poor outcome in gastric cancer. These patients generally have a prognosis similar to patients who are clinically or radiologically classified as having Stage IV disease. Similar, although fewer, observations have been made in patients with pancreatic cancer. If identified prior to scheduled resection, an extensive operation may not be required. The purpose of this pilot trial is to investigate the ability of a quantitative RT-PCR assay to detect cancer cells in peritoneal washings of patients undergoing laparoscopy for gastric or pancreatic cancer. This assay may detect mRNA overly expressed in gastric or pancreatic cancer patients with malignant cells in the peritoneum which cannot be detected by less sensitive means. Results of this assay will be compared to cytology results, as detected by standard Papanicolaou staining, during routine laparoscopic peritoneal washings in the absence of visible M1 disease. We anticipate enrolling 50 gastric cancer patients and 50 pancreatic cancer patients who will be undergoing laparoscopy as part of their initial management. We plan to enroll 30 patients undergoing laparoscopy for a presumed benign condition (e.g., gallstones, prophylactic bilateral salpingo-oophorectomy [BSO]) as negative controls. We estimate accrual will take approximately 12 months. Once this assay is established with this pilot study, we plan to evaluate prospectively the incidence, predictors, and clinical significance of positive cytology, as detected by standard Papanicolaou stainingand RT-PCR of tumor markers. This study does not conflict with any existing protocol at Memorial Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age and older.
* Presentation of gastric or pancreatic cancer based on objective findings on at least one of: CT scan; endoscopy; pathologic examination.
* Informed consent, indicating the investigational nature of this study in keeping with the policies of Memorial Sloan-Kettering Cancer Center.
* For negative controls, any patient undergoing a laparoscopy for presumed benign disease (e.g., cholecystectomy, hernia repair, BSO)

Exclusion Criteria:

* Under 18 years of age.
* Inability to speak or read English, and an appropriate translator is not identifiable.
* Unable or unwilling to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be those with a diagnosis of gastric or pancreatic cancer who present to the Surgical Services at Memorial Sloan-Kettering Cancer Center, who are candidates for surgical treatment, and are scheduled for laparoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of this pilot trial is to investigate the ability of quantitative RT-PCR to detect cancer cells in peritoneal washings of patients undergoing laparoscopy for gastric or pancreatic cancer. | conclusion of study

SECONDARY OUTCOMES:
The secondary objective of this pilot study is to estimate the sensitivity, specificity, false positive, and false negative rate of peritoneal cancer cell detection by quantitative RT-PCR. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Coit, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center website — http://www.mskcc.org